CLINICAL TRIAL: NCT03656120
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase Ⅱb Clinical Trial of Thienorphine Hydrochloride Tablets for the Efficacy, Safety, and Optimal Dosing of Relapse Prevention After Opioid Dependence Detoxification
Brief Title: A Study of Thienorphine Hydrochloride Tablets in Relapse Prevention Treatment of Opioid Dependence
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wei Hao (Other)
Collaborators: Beijing ziduhongye technology development co. LTD (Unknown); Institute of Pharmacology and Toxicology, Academy of Military Medical Science (Unknown); Shanghai Mental Health Center (Other); West China Hospital (Other); Wuhan Mental Health Centre (Other)
Responsible Party: Sponsor-Investigator, Wei Hao, Deputy Director, Institute of Mental Health, Second Xiangya Hospital, Central South University, Central South University
Organization: Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 100000-068945
Record Dates: First submitted 2018-08-29; First posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Opioid Dependence
Keywords: opioid dependence; thienorphine hydrochloride
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.2mg group (Experimental): Participants are taking 0.2mg thienorphine hydrochloride table once a day for 12 weeks.
  Interventions: Drug: 0.2mg group
- 0.5mg group (Experimental): Participants are taking 0.5mg thienorphine hydrochloride table once a day for 12 weeks.
  Interventions: Drug: 0.5mg group
- placebo control group (Placebo Comparator): Participants only taking placebo once a day for 12 weeks.
  Interventions: Drug: placebo control group

INTERVENTIONS:
Drug: 0.2mg group — Thienorphine hydrochloride dose was set as 0.2mg per day,last for 12 weeks.
  Arms: 0.2mg group
Drug: 0.5mg group — Thienorphine hydrochloride dose was set as 0.2mg per day for the first week and increased to 0.5mg per day from the second week, last for 11 weeks.
  Arms: 0.5mg group
Drug: placebo control group — Participants only take placebos for 12 weeks during the research.
  Arms: placebo control group

SUMMARY:
Opioid addiction is common worldwide. Thienorphine hydrochloride is a newly partial opioid receptor agonist drugs. It's affinity with opioid receptors was much higher than opioids, which could effectively prevents opioid dependence by stop opioids competition for opioid receptors and causing opioid dependence. The aim of this research was to determine whether thienorphine hydrochloride would reduce opioid use and better preventing relapse among opioid addicts.

DETAILED DESCRIPTION:
Opioids dependence is a chronic brain disease, with a much higher rate of relapse rate. Relapse prevention is important for opioid dependence treatment. Thienorphine hydrochloride, derivatives of buprenorphine, is one of the receptor partial agonists. Previous research indicated that, it may be a safe and effective treatment for the prevention of opioid dependent patients after detoxification. In this multicenter, randomized, double-blind, placebo-controlled, phase Ⅱb clinical trial, we are aimed to evaluate the efficacy of thienorphine hydrochloride tablets for anti-relapse therapy after opioid dependence detoxification treatment, determining the optimal dose of thienorphine hydrochloride tablets, and further evaluate the safety of thienorphine hydrochloride for patients with opioid dependence. 180 eligible patients are going to be recruited and randomly assigned to 0.2mg/day group, 0.5mg/day group and placebo control group after they provided their consent forms. Subjects in each group would receive assigned treatment for 12 weeks. Primary outcome measure was retention time of each participants during these 12 weeks. Urine test for opioids, changing of withdrawal score and craving, self-reported euphoria after using heroin, subjects and researchers' overall evaluation of treatment efficacy are secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Currently meets the diagnostic criteria for DSM-IV opioid dependence, with a history of opioids using more than 1 year; having relapsed for opioids for at least twice, and meets one of the following criterion:

   1.1 Opioid dependent patients (including heroin dependent patients or patients undergoing methadone maintenance treatment) treated with buprenorphine and meeting the following criteria: 1.1.1 Taking buprenorphine 2 mg per day for at least 3 consecutive days; 1.1.2 Clinical Opioid Withdrawal Symptom Scale (COWS) score ≤ 4; 1.1.3 Negative urine test results for morphine and methadone; 1.2 Having been stopped to using opioids. Negative urine test results for morphine, methadone and buprenorphine. As well as negative result for naloxone-precipitated tests ((including patients returning to the community from drug rehabilitation agencies).
2. Age 18 to 60 years old, male and female
3. Weight 40 ~ 95kg
4. Able to communicate with researchers, willing to receive anti-relapse therapy, and provide signed consent forms.

Exclusion Criteria:

1. Substance dependence other than nicotine;
2. Severe psychiatric disorders;
3. Severe physical illnesses, including severe digestive, cardiovascular, respiratory, and endocrine systems problems;
4. Patients with severe chronic pain;
5. Women in pregnancy or lactation
6. Patients who do not have effective contraception methods
7. Systolic/diastolic pressure is higher than 150/100mmHg or lower than 85/60mmHg
8. Heart rate <50 beats / min;
9. Severe liver or kidney dysfunction or severe abnormalities confirmed by laboratory test (liver function indicators ALT, AST are more than 3 times higher than the upper limit of normal values; any of the renal function indicators BUN, Cr that is higher than the upper limit of normal 1.5 times and above);
10. Allergic to buprenorphine or other similar drugs;
11. Patients with dysuria or urinary retention symptoms;
12. People with severe habitual constipation;
13. Those with HIV infection;
14. Poor adherence;
15. Participants enrolled in other clinical trials within 4 weeks prior to enrollment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-08-31 (Estimated); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
days of retention in outpatient treatment | up to 12 weeks
  Primary outcome measure was retention time of each participants during these 12 weeks, defined as from the beginning of randomized into assigned group to the days participants decided to quit the research for the following reasons: (1) Subjects were not receiving assigned therapy for seven consecutive days or more; (2) the subject cannot continue to participate in the study for other reasons; (3) The researchers decided that the subject should stop the study based on their clinical diagnosis and treatment; (4) subjects withdrew their consent form.

SECONDARY OUTCOMES:
opioids negative rate through urine test | up to 12 weeks
  For each subject，opioids negative rate was defined as the number of negative urine test during the 12-week treatment divided by the number of urine tests each subject should performed at the end of the study. Missed test is treated positively by urine test.
Change of withdrawal score of Clinical Opioid Withdrawal Symptom Scale (COWS) from baseline to 12 weeks | up to 12 weeks
  Clinical Opioid Withdrawal Symptom Scale (COWS) is calculates as the change in the subject's COWS score over the 12-week period compared to baseline. COWS scale contains a total of 32 items, and the contents of the item basically cover all symptoms and signs of opioid withdrawal. Each symptom is divided into four levels, ranging from 0 (no symptoms at all) to 3 (severe symptoms).
Change of craving from baseline in Visual Analog Scale (VAS) at 12 weeks | up to 12 weeks
  A 10-point Visual Analog Scale (VAS) was used to assess subjective self-report craving for opioids, where the subject was asked to quantify his/her subjective state of craving for opioids by marking a point on a line which is anchored at one end by words describing an absence of the subjective craving state (0 point) and at the other end by words describing a maximal intensity of craving state (10 points).
Change of self-reported euphoria after using heroin | up to 12 weeks
  Within these 12 weeks, euphoria scores of subject lapsed to heroin are collect if the subject lapsed to heroin.
Subjects ' overall evaluation of efficacy of relapse prevention treatment of thienorphine hydrochloride tablets | up to 12 weeks
  At the end of the 12-week study, subjects are going to evaluate the overall treatment efficacy of thienorphine hydrochloride during these 12-week period using a five-point scale. The scale is divided into 5 levels: very good, good, fair, poor, and very poor.
Researchers' overall evaluation of efficacy of relapse prevention treatment of thienorphine hydrochloride tablets | up to 12 weeks
  At the end of the 12-week study, researchers are going to evaluate the overall treatment efficacy of thienorphine hydrochloride during these 12-week period using a five-point scale. The scale is divided into 5 levels: very good, good, fair, poor, and very poor.

CONTACTS AND LOCATIONS:
Overall Officials: Weri Hao, Doctor, Principal Investigator — The Second Xiangya Hospital，Central South University, Changsha, China